CLINICAL TRIAL: NCT05500495
Title: The Association Between Doppler Parameters of Superior Mesenteric Artery(SMA) and Prolonged Mechanical Ventilation(PMV) in Patients After Cardiac Valve Surgery
Brief Title: The Association Between Intestinal Perfusion and Prolonged Mechanical Ventilation in Patients After Cardiac Valve Surgery
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-3088
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Patient After Cardiac Valve Surgery; Patient With Prolonged Mechanical Ventilation
Keywords: Pulsatility index of the superior mesenteric artery; Prolonged Mechanical Ventilation; cardiac valve surgery; intestinal perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prolonged mechanical ventilation group: patients had 96 hours or more (PMV group).
  Interventions: Other: no intervention
- control group: patients had less than 96 hours of mechanical ventilation (control group)
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Background This study aimed to confirm that alterations in Doppler parameters of superior mesenteric artery(SMA) blood flow caused by intestinal hypoperfusion are associated with prolonged mechanical ventilation(PMV) in patients after cardiac valve surgery.

Methods The patients' basic hemodynamics parameters, and the SMA blood flow parameters monitored by Doppler ultrasound were collected in the supine position at admission. The length of mechanical ventilation continued to be monitored. The SMA Doppler parameters were measured again when the patient was extubated. PMV was defined as MV≥96 hours.

DETAILED DESCRIPTION:
Patient enrollment This prospective observational study was performed in the 15-bed adult critical care unit in Adult General Hospital from January 2021 to March 2022.

The inclusion criteria were as follows: 1) patients admitted to ICU immediately after cardiac valve surgery; 2) age 18-80 years; 3) sinus rhythm; 4) without active bleeding or pneumothorax, and 5) complete measurement data.

The exclusion criteria were as follows: 1) history of peripheral vascular disease, 2) patients with severe stenosis defined as SMA peak systolic velocity (SMA-PSV >275 cm/s or SMA-PSV/abdominal aorta peak velocity of >3, 3) hepatic dysfunction or liver cirrhosis, portal hypertension, 4) cancer or end-stage renal diseases, 5) poor quality of abdominal ultrasound images.

Doppler ultrasound monitoring Doppler ultrasound was performed with an ultrasound system consisting of a 2-5 MHz C60xp Probe (X-Porte Ultrasound System, FUJIFILM SONOSITE, INC., USA). Blood flow parameters were measured by two physicians, each physician measured twice and averaged, and then averaged the two results. Each of the two ICU physicians had more than four years of experience in critical ultrasound and obtained certification from the Chinese Critical Ultrasound Study Group. Two skilled physicians conducted a total of 40 measurements on ten patients after cardiac valve surgery to evaluate inter-observer reproducibility.

The SMA flow was measured 1 cm proximal to the abdominal aorta. The angle of insonation was < 60°. The time-velocity waveform readings were used to measure the peak systolic velocity (PSV), end-diastolic velocity(EDV), resistance index(RI), time-averaged mean velocity(TAMV), pulsatility index (PI), according to the calculation software carried by the ultrasound. PI=(PSV-EDV)/TAMV, and RI=(PSV-EDV)/PSV.

Data collection Demographic information was recorded for further analyses (e.g., age, gender, EuroSCORE-II, sequential organ failure assessment (SOFA) score, body mass index (BMI), and hemodynamic parameters and blood gas analysis data). In addition, types of operation and operation time were collected. Moreover, outcome variables (e.g., hospital mortality, time of MV, length of ICU stay) were recorded for further comparison.

Statistical analysis The median plus the interquartile range (IQR) or mean standard deviation is used to show demographic data. The Shapiro-Wilk test was used to evaluate normality. The differences between groups were compared using the student's t-test for continuous variables with normality distribution and the Mann-Whitney U test for those without normality distribution. The differences between groups for categorical variables were compared by performing a Chi-square test. Correlations between variables and PMV were assessed by conducting logistic regression analysis. Variables showing statistical significance in the univariate logistic regression were selected covered in the multivariate logistic regression. Furthermore, to evaluate the predictive ability of the variables for PMV, a receiver operating characteristic (ROC) curve was applied. Statistical significance was set at P < 0.05. All analyzed P-values were two-sided. Statistical analyses were performed using the SPSS 25.0 software package (SPSS, Chicago). Bland-Altman plots with the mean difference and 95 percent limit of agreement (LOA) were used to assess inter-observer agreement, and statistical analyses were done using MedCalc Statistical software.

ELIGIBILITY:
Inclusion Criteria:

1) patients admitted to ICU immediately after cardiac valve surgery; 2) age 18-80 years; 3) sinus rhythm; 4) without active bleeding or pneumothorax, and 5) complete measurement data.

Exclusion Criteria:

1) history of peripheral vascular disease, 2) patients with severe stenosis defined as SMA peak systolic velocity (SMA-PSV >275 cm/s or SMA-PSV/abdominal aorta peak velocity of >310, 3) hepatic dysfunction or liver cirrhosis, portal hypertension, 4) cancer or end-stage renal diseases, 5) poor quality of abdominal ultrasound images.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient was enrolled in the 15-bed adult critical care unit in Adult General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
hours of mechanical ventilation | within 30mins at ICU admission
  hours of mechanical ventilation

SECONDARY OUTCOMES:
ICU residence time | within 30mins at ICU admission
  ICU residence time

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No